CLINICAL TRIAL: NCT02662946
Title: Evaluation of Intestinal Vascolarization by Intraoperative Angiography With Indocianine Green During Laparoscopi Rectal Resection or Left Colectomy: Predictive Value on Anastomotic Leak.
Brief Title: Evaluation of Intestinal Vascolarization With Indocianine Green Angiography During Rectal Resection or Left Colectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Paola De Nardi, MD, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Angio-Co-Re
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Rectal Disease; Sigmoid Disease
MeSH Terms: conditions — Rectal Diseases; Sigmoid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICG- angiography (Experimental): Colonic resection margins and colo-rectal anastomosis are intraoperatively assessed using fluorescence angiography to evaluate colonic perfusion. If perfusion at the resection margin is judged "insufficient" the colon is re-resected to obtain a satisfactory perfusion
  Interventions: Procedure: ICG- angiography
- No angiography (Active Comparator): Subjective measures are employed to determine anastomotic perfusion
  Interventions: Procedure: No angiography

INTERVENTIONS:
Procedure: ICG- angiography — Angiography with ICG prior to and after anastomosis. Extension of colon resection based on ICG angiography results
  Arms: ICG- angiography
Procedure: No angiography — Extension of resection based on subjective measures
  Arms: No angiography

SUMMARY:
A randomized controlled multicenter trial on the usefulness of intraoperative angiography with indocyanine green to assess anastomosis perfusion in patients who undergo laparoscopic rectal resection or left colectomy.

DETAILED DESCRIPTION:
Anastomotic leakage after colorectal surgery is a severe complication. One possible cause of anastomotic leakage is insufficient vascular supply. The aim of this study is to evaluate the usefulness of intraoperative assessment of vascular anastomotic perfusion in laparoscopic colorectal surgery using indocyanine green (ICG)-enhanced fluorescence, in order to assess if the information of the ICG angiography could lead to change the site of resection and improving the anastomotic leak rate. Two-hundred and eight patients, undergoing rectal resection or left colectomy, for benign or malignant disease, with high vessels ligation, will be randomized intro 2 arms: ICH angiography (colonic perfusion is intraoperatively assed with ICG angiography and level of resection is selected based on the fluorescence) and Control (resection is performed with subjective judgment). The rate of postoperative leak in the two groups will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult patiens
* laparoscopic rectal resection or left colectomy

Exclusion Criteria:

* rectal amputation
* no anastomosis
* allergy to iodine or indocyanine green

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paola De Nardi, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Nardi P, Elmore U, Maggi G, Maggiore R, Boni L, Cassinotti E, Fumagalli U, Gardani M, De Pascale S, Parise P, Vignali A, Rosati R. Intraoperative angiography with indocyanine green to assess anastomosis perfusion in patients undergoing laparoscopic colorectal resection: results of a multicenter randomized controlled trial. Surg Endosc. 2020 Jan;34(1):53-60. doi: 10.1007/s00464-019-06730-0. Epub 2019 Mar 21. PMID 30903276